CLINICAL TRIAL: NCT01548287
Title: A Phase IIa Safety and Tolerability Study to Investigate the Effect on Sleep of 3 Doses of AZD5213 and Placebo in Patients With Mild Alzheimer's Disease and Mild Cognitive Impairment During 4 Weeks of Treatment, Placebo-Controlled
Brief Title: A Study of the Safety and Tolerability of AZD5213 Effect on Sleep for Patients With Alzheimer's/Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3030C00005
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Mild Cognitive Impairment; Mild Alzheimer's Disease
Keywords: Mild Cognitive Impairment; Mild Alzheimer's disease; Safety; Tolerability
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD5213 doseA (Experimental): AZD5213 doseA daily
  Interventions: Drug: AZD5213
- AZD5213 doseB (Experimental): AZD 5213 doseB daily
  Interventions: Drug: AZD5213
- AZD5213 doseC (Experimental): AZD5213 doseC daily
  Interventions: Drug: AZD5213
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD5213 — AZD5213 doseA daily
  Arms: AZD5213 doseA
Drug: AZD5213 — AZD5213 doseB daily
  Arms: AZD5213 doseB
Drug: AZD5213 — AZD5213 doseC daily
  Arms: AZD5213 doseC
Other: Placebo — Placebo tablet daily
  Arms: Placebo

SUMMARY:
This is a study where AZD5213 or placebo is given to patients with Mild Alzheimer's Disease or Mild Cognitive Impairment in a blinded and random assignment. The main study objective is to estimate the relationship of sleep duration versus dose after 4 weeks of treatment.

DETAILED DESCRIPTION:
A Phase IIa Safety and Tolerability Study to Investigate the Effect on Sleep of 3 Doses of AZD5213 and Placebo in Patients with Mild Alzheimer's Disease and Mild Cognitive Impairment During 4 Weeks of Treatment, Designed as a Randomized, Double-Blind, Multi-Center, Parallel Group, Placebo-Controlled Study

ELIGIBILITY:
Inclusion Criteria:

* Patient and study partner to sign informed consent before initiation of any study-related procedures.
* Clinical diagnosis of Alzheimers (AD) or mild cognitive impairment (MCI) disease.
* Single caregiver for at least 6 months prior to Screening, capable of accompanying the patient on clinic visits as needed. The caregiver must either be living with or visiting the patient at least 10 hours per week, split over multiple (at least 2) days, for the duration of the study.
* Single study partner, for at least several months prior to Screening, capable of accompanying the patient on clinic visits as needed. The study partner must either be living with or visiting the patient at least 3 days per week for the duration of the study.
* A body mass index (BMI=weight/height2) of 18 kg/m2 to 32 kg/m2.

Exclusion Criteria:

* Significant neurological disease or dementia other than AD or MCI.
* Current episode or symptoms of major depressive disorder or other major psychiatric disorder.
* History of self-reported sleep duration of less than 4 hours per night or less than 4 hours average total sleep time per night during Baseline PSG assessment.
* History or present symptoms of a sleeping disorder such as sleep apnea.
* History of cancer in the last 5 years.
* Use of anti-AD drugs (including off-label drugs and herbal medications) with the exception of donepezil, memantine, and/or rivastigmine transdermal system, as monotherapy or in combination in the following conditions: treatment with donepezil (5 mg to 10 mg daily), memantine, and/or rivastigmine transdermal system or combination regimens for at least 3 months and a stable dose(s) for the last 2 months prior to randomization is allowed.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Alexander, MD, Study Director — AstraZeneca Research & Development, Neuroscience iMed, 141 Portland Street, Cambridge, MA 02139; Roza Hayduk, MD, Study Director — Quintiles 10201 Wateridge Circle San Diego, CA
Locations (13):
- United States (13):
  - Research Site, Phoenix, Arizona
  - Research Site, Indio, California
  - Research Site, Lomita, California
  - Research Site, San Francisco, California
  - Research Site, Delray Beach, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Eatontown, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Salt Lake City, Utah

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- See also: D3030C00005_Clinical_Study_Report_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1316&filename=D3030C00005_Clinical_Study_Report_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 164 subjects signed informed consent and 83 failed to qualify at the first screening visit for participation in the study.
Groups:
- AZD5213 Dose A: AZD5213 AZD 0.5 mg daily
- AZD5213 Dose B: AZD 5213 2.0 mg daily
- AZD5213 Dose C: AZD5213 6.0 mg daily
- Screening Only: Screening period only, not randomized
Period: Screening
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo | Screening Only
Started | 19 | 22 | 20 | 20 | 83
Completed | 19 | 22 | 20 | 20 | 0
Not Completed | 0 | 0 | 0 | 0 | 83
Not completed — No reason provided | 0 | 0 | 0 | 0 | 9
Not completed — Did not meet eligibility criteria | 0 | 0 | 0 | 0 | 74
Period: Randomized Period
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo | Screening Only
Started | 19 | 22 | 20 | 20 | 0
Completed | 19 | 20 | 13 | 20 | 0
Not Completed | 0 | 2 | 7 | 0 | 0
Not completed — Did not meet inclusion criteria | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo | Total
Number analyzed (Participants) | 19 | 22 | 20 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (8.02) | 65.1 (8.04) | 69.3 (10.32) | 64.2 (7.62) | 66.1 (8.62)
Gender [Count of Participants; unit: Participants]
  Female | 12 | 16 | 13 | 15 | 56
  Male | 7 | 6 | 7 | 5 | 25
Mini-Mental State Examination [Mean (Standard Deviation); unit: Scores on scale] — Mini-Mental Scale Examination, Total Score range 0-30, higher score indicates less cognitive impairment
  Scores on scale | 27.2 (1.38) | 27.0 (2.01) | 26.1 (1.62) | 27.0 (1.88) | 26.8 (1.77)
Alzheimers disease (AD)/Mild cognitive impairment (MCI) [Number; unit: Participants]
  AD | 3 | 6 | 5 | 5 | 19
  MCI | 16 | 16 | 15 | 15 | 62
Concomitant donepezil administration [Number; unit: Participants]
  Yes | 2 | 1 | 3 | 3 | 9
  No | 17 | 21 | 17 | 17 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Sleep Time (TST) After 4 Weeks of Treatment, Based on PSG Measurement.
Description: Total sleep time (TST) is defined as the total time in minutes, that subjects were determined to be in a sleep state by polysomnography (PSG) measurement.
Time Frame: Baseline and Week 4.
Population: Primary analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Minutes
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Number analyzed (Participants) | 19 | 20 | 13 | 20
Minutes | 6.43 [-12.74 to 25.61] | -12.53 [-31.32 to 6.27] | -19.41 [-41.91 to 3.08] | 14.48 [-4.31 to 33.27]

2. Secondary Outcome: Change From Baseline in Sleep Efficiency After 4 Weeks of Treatment, Based on PSG Measurements.
Time Frame: Baseline and Week 4.
Population: Primary analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: % change
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Number analyzed (Participants) | 19 | 20 | 13 | 20
% change | 0.08 [-3.15 to 3.32] | -1.51 [-4.68 to 1.66] | -2.82 [-6.61 to 0.97] | 0.96 [-2.20 to 4.13]

3. Secondary Outcome: Change From Baseline in Latency to Persistent Sleep After 4 Weeks of Treatment, Based on PSG Measurements.
Time Frame: Baseline and Week 4.
Population: Primary analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Rank transformed duration (minutes)
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Number analyzed (Participants) | 19 | 20 | 13 | 20
Rank transformed duration (minutes) | -2.23 [-18.44 to 13.98] | 14.48 [-1.34 to 30.31] | -5.84 [-24.91 to 13.23] | -5.68 [-21.54 to 10.18]

4. Secondary Outcome: Change From Baseline in Night Total Sleep Time After 4 Weeks of Treatment, Based on Actigraphy Recording.
Description: Change from baseline in night total sleep time after 4 weeks of treatment: assessed if valid baseline and week 4 actigraphy data
Time Frame: Baseline and Week 4.
Population: Subset of Primary Analysis Set with valid actigraphy data
Measure: Least Squares Mean (90% Confidence Interval); unit: Minutes
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Number analyzed (Participants) | 17 | 19 | 11 | 17
Minutes | 7.07 [-14.88 to 29.02] | -12.42 [-34.92 to 10.07] | -18.97 [-45.96 to 8.02] | -7.51 [-29.47 to 14.44]

5. Secondary Outcome: Change From Baseline in Latency of Persistent Sleep After 4 Weeks of Treatment, Based on Actigraphy Recording.
Description: Change from baseline in latency of persistent sleep after 4 weeks of treatment, based on participants with valid baseline and week 4 actigraphy data
Time Frame: Baseline and Week 4.
Population: Subset of Primary Analysis Set with valid actigraphy data
Measure: Least Squares Mean (90% Confidence Interval); unit: Minutes
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Number analyzed (Participants) | 17 | 19 | 11 | 17
Minutes | 1.77 [-5.41 to 8.96] | 9.84 [2.86 to 16.81] | -6.85 [-15.50 to 1.81] | 2.70 [-4.65 to 10.06]

6. Secondary Outcome: Change From Baseline in Sleep Efficiency After 4 Weeks of Treatment, Based on Actigraphy Recording.
Description: Change from baseline in sleep efficiency after 4 weeks of treatment, based on participants with valid baseline and week 4 actigraphy data
Time Frame: Baseline and Week 4.
Population: Subset of Primary Analysis Population with valid actigraphy data
Measure: Least Squares Mean (90% Confidence Interval); unit: % (efficiency=% of time asleep)
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Number analyzed (Participants) | 17 | 19 | 11 | 17
% (efficiency=% of time asleep) | -0.05 [-3.65 to 3.55] | -3.20 [-6.69 to 0.30] | -1.92 [-6.20 to 2.35] | -1.83 [-5.46 to 1.80]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the follow-up (up to 38 days total)
Arm/Group | AZD5213 Dose A | AZD5213 Dose B | AZD5213 Dose C | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22 | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/19 | 11/22 | 13/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD5213 Dose A (N=19) | AZD5213 Dose B (N=22) | AZD5213 Dose C (N=20) | Placebo (N=20)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD5213 Dose A (N=19) | AZD5213 Dose B (N=22) | AZD5213 Dose C (N=20) | Placebo (N=20)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 8 (9) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoasthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypnagogic hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days